CLINICAL TRIAL: NCT04463121
Title: Pressure-Volume (PV) Measurements for Evaluating the Changes in the Ventricular Preload and Autonomic Nervous System Using BackBeat Medical Cardiac Neuromodulation Therapy (CNT) Signals in an Acute Study
Brief Title: Preload and Autonomic Responses With Cardiac Neuromodulation Therapy (CNT) (CS-06)
Acronym: CS-06
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BackBeat Medical Inc (Industry)
Collaborators: CD Leycom (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BBM MOD PV CS-06
Record Dates: First submitted 2020-06-30; First posted 2020-07-09 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Bradycardia; Hypertension, Systolic
MeSH Terms: conditions — Bradycardia; Isolated Systolic Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute CNT pacing signals testing (Experimental): Acute study procedure will be carried out prior to a pacemaker implantation or replacement: pacemaker Right Atrial (RA) and Right Ventricular (RV) leads will be positioned according to standard procedure for pacemaker implant and connected to a Moderato® System IPG, via a single use, sterile Pacing System Analyzer (PSA) cable. The Moderato IPG will deliver CNT signals.
  Furthermore, a standard conductance catheter in the left ventricle will measure cardiac volumes and pressure. Arterial blood pressure will be obtained as well.
  A range of CNT signal parameters will be used to assess the effect on sympathetic activity at different positions of the RV pacing lead while ventricular pressure and volume and arteial pressure signals will be assesed for cardiac function, sympathetic activity and blood pressure. The effects of CNT signal over a range of parameter settings will be studied for the different RV lead positions.
  Interventions: Device: Moderato IPG's CNT pacing signals; Device: CD Leycom Pressure/Volume Combination Catheters

INTERVENTIONS:
Device: Moderato IPG's CNT pacing signals — Assesment of cardiac function and sympatheric activity will be obtained simultaneously
Device: CD Leycom Pressure/Volume Combination Catheters — Simultaneous recording of the Pressure, Volume measurements and ECG signals will be done for constant monitoring of intra-ventricular pressure and volume.

SUMMARY:
This investigation will evaluate the effect of RV pacing lead position on cardiac function and the modulation of the autonomic nervous system with Cardiac Neuromodulation Therapy (CNT) pacing signals. The study will be performed acutely prior to a pacemaker implant.

DETAILED DESCRIPTION:
Subjects indicated for a dual chamber pacemaker implant or replacement who are not 100% dependent on right ventricular pacing may be eligible to participate in the study.

This investigation will evaluate the effect of RV pacing lead position on cardiac function and the modulation of the autonomic nervous system using Cardiac Neuromodulation Therapy (CNT) pacing signals at different positions of the RV pacing lead.

A standard conductance catheter will be introduced through the femoral artery and advanced into the left ventricle to measure cardiac volumes and pressure.

Arterial blood pressure will be measured from the other femoral artery with an additional sheath.

The Moderato® IPG will be used to generate Cardiac Neuromodulation Therapy (CNT) signals and deliver them to the patient through the cable and leads. A range of CNT signal parameters will be used to assess the effect on sympathetic activity at different positions of the RV pacing lead. Ventricular pressure and volume readings from the conductance catheter and arterial pressure readings will be recorded and analyzed to assess the effect of CNT signals on cardiac function, sympathetic activity and blood pressure.

The effects of CNT signal over a range of parameter settings will be studied for the different RV lead positions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age
2. Subject requires implantation or replacement of a dual chamber pacemaker or requires an upgrade from a single chamber to a dual chamber pacemaker
3. Subject has known Hypertension
4. Subject is willing and able to comply with the study and procedures.

Exclusion Criteria:

1. Subject has symptoms of heart failure, NYHA Class II or greater
2. Subject has significant (>2+) mitral regurgitation, aortic regurgitation or aortic stenosis.
3. Subject has permanent atrial fibrillation
4. Subject has atrial fibrillation on the day of the study.
5. Subject has hypertrophic cardiomyopathy, restrictive cardiomyopathy or interventricular septal thickness ≥15 mm
6. Subject is on dialysis
7. Subject has a history of prior neurological events (stroke or TIA) within the past year or a neurological event (stroke or TIA) at any prior time that has resulted in residual neurologic deficit.
8. Subject has a history of autonomic dysfunction
9. Women who are pregnant or breast-feeding
10. Subject cannot or is unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Effects of the Moderato CNT pacing signals on cardiac function | approximately one hour
  Left ventricular pressure (mmHg) and Volume (ml) will be obtained by a multisensor catheter which provides real-time, beat-to-beat intra-ventricular measurement of cardiac function and performance. Data will be used to generate Pressure-Volume Loops, an aknowledged way to describe hemodynamic changes. CNT signals (alternating short and long atrioventicular sequences 40-150 ms) will be delivered at the same by right ventricular pacemaker leads temporarely connected to the Moderato device.
Effects of CNT pacing signals on blood pressure | aproximately onr hour
  Blood pressure (mmHg) will be obtained in parallel with a Millar catheter from the femoral artery througout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, PhD, Principal Investigator — Na Homolce Hospital
Locations (1):
- Na Homolce Hospital, Prague, Czechia

REFERENCES:
- [Background] Yang B, Wang Y, Zhang F, Ju W, Chen H, Mika Y, Aviv R, Evans SJ, Burkhoff D, Wang J, Chen M. Rationale and evidence for the development of a durable device-based cardiac neuromodulation therapy for hypertension. J Am Soc Hypertens. 2018 May;12(5):381-391. doi: 10.1016/j.jash.2018.03.004. Epub 2018 Mar 21. PMID 29628351
- [Background] Neuzil P, Merkely B, Erglis A, Marinskis G, de Groot JR, Schmidinger H, Rodriguez Venegas M, Voskuil M, Sturmberger T, Petru J, Jongejan N, Aichinger J, Kamzola G, Aidietis A, Geller L, Mraz T, Osztheimer I, Mika Y, Evans S, Burkhoff D, Kuck KH; BackBeat Study Investigators. Pacemaker-Mediated Programmable Hypertension Control Therapy. J Am Heart Assoc. 2017 Dec 23;6(12):e006974. doi: 10.1161/JAHA.117.006974. PMID 29275370
- [Background] de Roest GJ, Allaart CP, Kleijn SA, Delnoy PP, Wu L, Hendriks ML, Bronzwaer JG, van Rossum AC, de Cock CC. Prediction of long-term outcome of cardiac resynchronization therapy by acute pressure-volume loop measurements. Eur J Heart Fail. 2013 Mar;15(3):299-307. doi: 10.1093/eurjhf/hfs190. Epub 2012 Nov 25. PMID 23183349